CLINICAL TRIAL: NCT04741438
Title: A Randomised, Comparative, Prospective, Multicentre Study of the Efficacy of Nivolumab + Ipilimumab Versus Pazopanib Alone in Patients With Metastatic or Unresectable Advanced Sarcoma of Rare Subtype (RAR-Immune)
Brief Title: Efficacy of the Combination of Nivolumab and Ipilimumab as a Treatment in Patients With Sarcoma of Rare Subtype
Acronym: RAR-Immune
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET 20-128_RAR-IMMUNE
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Sarcoma
Keywords: Sarcoma of rare subtype; Metastatic sarcoma; Unresectable advanced sarcoma; Nivolumab; Ipilimumab; Randomization; Pazopanib; Progression free-survival; Best Overall Response; Objective response rate; Duration of response; Time to treatment failure; Overall survival; Quality of Life; Tolerance profile
MeSH Terms: conditions — Sarcoma | interventions — Nivolumab; Ipilimumab; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Arm A (Experimental arm).
  * Nivolumab 3 mg/kg
  * Ipilimumab 1 mg/kg
  Interventions: Drug: Nivolumab and IPILIMUMAB
- Arm B (Active Comparator): Arm B (Control arm). Pazopanib 800 mg/day
  Interventions: Drug: Pazopanib Oral Tablet [Votrient]

INTERVENTIONS:
Drug: Nivolumab and IPILIMUMAB — The combination of Nivolumab+Ipilimumab will be given to patients as follows:
  * Nivolumab: 3 mg/kg IV over 30 minutes every 2 weeks for 4 cycles.
  * Ipilimumab 1 mg/kg IV over 60 minutes every 6 weeks for 4 cycles. After completion of 4 courses with ipilimumab, patients continue receiving nivolumab IV at the dose of 480 mg Q4W in the absence of disease progression or unacceptable toxicity for a maximum of 18 months.
  Nota Bene: A cycle is defined as a 6-weeks period.
  The planned treatment period is 24 months
  Nivolumab and Ipilimumab must be injected the same day every 6 weeks (Q6W). In case of toxicity, dose will be delayed, but will not be reduced.
  Arms: Arm A
Drug: Pazopanib Oral Tablet [Votrient] — Treatment by pazopanib 800 mg/day per os, continuously during a maximum 24 months.
  In case of toxicity, dose will be delayed and reduced.
  Arms: Arm B

SUMMARY:
This is a randomized open label study, with 2 arms treatments conducted in patients with metastatic or unresectable advanced sarcoma of rare subtype; previously treated by anthracycline-based regimen except for whom standard therapy does not exist or is not considered appropriate by the Investigator.

In the experimental arm, patients will receive the combination of Nivolumab + Ipilimumab for a maximum of 24 months, whereas in the control arm, patients will receive Pazopanib alone.

The purpose of the study is to know if the combination of nivolumab + ipilimumab can be more efficient than Pazopanib in terms of Progression-Free Survival.

DETAILED DESCRIPTION:
This is a randomized open label, comparative, prospective, multicentre phase III study.

The patients who meet the eligibility criteria will be randomly assigned (1:1) into one of the following treatments groups:

* Experimental arm: Nivolumab + Ipilimumab (24 months maximum)
* Control arm: Pazopanib alone (24 months maximum)

A randomization procedure will be used to obtain a balanced distribution of stratifications factors:

* The number of previous lines of treatment in advanced/metastatic setting: ≤1 line or >1 line (a treatment line is defined as a treatment initiation whatever the reason)
* The lymphocytes count at baseline: <1 g/L or ≥1 g/L.

After their eligibility has been confirmed, patients will be treated with:

* The combination of Nivolumab + Ipilimumab for 4 cycles. After completion of 4 cycles with Ipilimumab, patients continue receiving nivolumab IV (480 mg Q4W) in the absence of disease progression or unacceptable toxicity. A cycle is defined as a 6-weeks period.
* Or Pazopanib until disease progression or unacceptable toxicity. The planned treatment duration in both arm is maximum 24 months.

After the completion of treatment, patients will be followed up within 30 days after the last study treatment administration. The survival and disease status will be updated for all patients at the time of the end of the study.

The overall end of the study will be the Last Patient Last Visit (LPLV), defined as the End Of Treatment (EOT) visit of the last active patient.

ELIGIBILITY:
Inclusion Criteria:

I1. Age ≥ 18 years at the day of consenting to the study;

I2. Only histologically confirmed sarcoma of rare subtype, defined as one of the following subtypes:

* Angiosarcoma (AS)
* Alveolar Soft Part Sarcoma (ASPS)
* Clear Cell Sarcoma (CCSA)
* Desmoplastic Small Round Cell Tumour (DSRCT)
* Sclerosing Epithelioid Fibrosarcoma (SEF)
* Perivascular Epithelioid Cell Tumour (PEComa)
* Intimal sarcoma (IS)
* Extraskeletal Myxoid Chondrosarcoma (EMC)
* Solitary Fibrous Tumour (SFT)
* Epithelioid HemangioEndothelioma (EHE)
* Inflammatory Myofibroblastic Tumour (IMT)
* Epithelioid sarcoma (ES)
* FibroSarcoma (FS)
* SMARCA-4 deficient sarcoma
* Malign Peripheral Nerve Sheath Tumours (MPNST)
* Chordoma;

I3. Metastatic disease or unresectable locally advanced malignancy that is resistant or refractory to standard therapy or for which standard therapy does not exist or is not considered appropriate by the Investigator;

I4. Measurable disease as per the RECIST version 1.1;

I5. Previously treated with anthracycline-based regimen except for whom standard therapy does not exist or is not considered appropriate by the Investigator: inclusion in first line is allowed (randomisation will be stratified according to the number of previous treatment lines);

I6. Performance Status (ECOG) of 0 or 1;

I7. Patients must have an adequate organ and bone marrow function at baseline;

* Absolute neutrophil count (ANC) ≥ 1.0 x 10 G/L
* Platelets ≥ 100 x 10 G/L
* Haemoglobin ≥ 9 g/dL (without transfusion within 7 days)
* Serum creatinine OR Calculated creatinine clearance as per MDRD or CKD-EPI formula ≤ 1.5 upper limit of normal (ULN) OR ≥ 40 mL/min /1.73m2
* Serum total bilirubin ≤ 1.5 ULN OR Direct bilirubin ≤ ULN for patients with total bilirubin levels > 1.5 ULN (except for patients with Gilbert disease for whom a total serum bilirubin ≤ 3ULN is acceptable).
* AST and ALT ≤ 3 ULN
* International Normalized Ratio (INR) and activated Partial Thromboplastin Time (aPTT) ≤ 1.5 ULN

I8. Women of childbearing potential must have a negative serum pregnancy test within 7 days before C1D1.

I9. Women of childbearing potential must agree to use 1 highly effective form of contraception from the time of the negative pregnancy test up to 3 months after the last dose of study drugs.

I10. Ability to understand and willingness for follow-up visits;

I11. Covered by a medical insurance;

I12. Signed and dated informed consent document indicating that the patient has been informed of all aspects of the trial prior to enrolment.

Exclusion Criteria:

E1. Concurrent use of any other approved or investigational antineoplastic agent;

E2. Prior or concurrent treatment with any antibody targeting PD1, PDL1, PDL2 or CTLA4;

E3. Prior treatment with pazopanib;

E4. Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.

Note:

* Asymptomatic patients with treated CNS lesions are eligible.
* Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy or surgery, with no need to repeat the screening brain scan;

E5. Patients using, or requirement to use while on the study, or not respecting the minimal wash-out period of medications listed below:

Forbidden concomitant medications and minimal wash-out period before Cycle 1 Day1

* Any approved anti-cancer systemic treatment including chemotherapy, hormonotherapy, biological therapy, or immunotherapy : 2 weeks
* Any investigational agents : 4 weeks
* Radiotherapy Note: palliative radiotherapy on non-target lesions is allowed. : 3 weeks
* Surgery
* Major surgical procedure, open biopsy, or significant traumatic injury : 4 weeks
* Abdominal surgery, abdominal interventions or significant abdominal traumatic injury : 60 days
* Live vaccines. Note: Influenza vaccination should be given during influenza season. Patients must not receive live attenuated influenza vaccine (e.g., FluMist®) : 4 weeks
* Systemic immunostimulatory agents, including but not limited to IFN-α, IFN-γ, or IL-2 : 4 weeks
* Immunosuppressive medication (including but not limited to corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) with the exceptions of intranasal, inhaled, or topical corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone (or 0.1mg/kg for pediatric patients), or an equivalent corticosteroid :2 weeks
* P-gp inhibitors : None
* Strong or moderate inhibitors of CYP3A4 : None
* Strong CYP3A4 inducers : None
* Oral or IV antibiotics :2 weeks

Note: Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection, pneumocystis or chronic obstructive pulmonary disease exacerbation) are eligible.

E6. History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis with the following exceptions:

* patients with a history of autoimmune-related hypothyroidism who are on stable thyroid replacement hormone therapy,
* patients with controlled Type 1 diabetes mellitus,
* patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are eligible provided that they meet the following conditions:

  * Rash must cover less than 10% of body surface area (BSA).
  * Disease is well controlled at baseline and only requiring low potency topical steroids.
  * No acute exacerbations of underlying condition within the previous 12 months requiring psoralen plus ultraviolet A radiation (PUVA), methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids;

E7. Patients with HIV, active B or C hepatitis infection, or any other active infection.

E8. Patients with active tuberculosis;

E9. Prior allogeneic bone marrow transplantation or solid organ transplant for another malignancy in the past;

E10. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan;

E11. Patients with a high-risk of hemorrhage or history of coagulopathy;

E12. Any contraindication to nivolumab, to ipilimumab or to pazopanib according to the Summary of Product Characteristics of each drug;

E13. History of other malignancy other than study disease (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix) unless the patient has been free of disease for at least 3 years;

E14. Patient under tutorship or curatorship or deprived of liberty;

E15. Pregnant or breast-feeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to 36 months
  The Progression-Free Survival defined as the time from the date of randomisation to the date of first documented progression or death due to any cause. Patients who have not progressed or died at the time of analysis will be censored at the time of the latest date of assessment.

SECONDARY OUTCOMES:
Best Overall Response (BOR) | up to 36 months
  The Best Overall Response will be defined as the best among all overall responses during the trial.
Objective Response Rate (ORR) | up to 36 months
  The Objective Response Rate will be defined as the proportion of patients with a best overall response of Complete Response (CR) or Partial Response (PR) during the trial.
Duration of Response (DOR) | up to 36 months
  in the patients whose BOR is either CR or PR, the DOR will be defined as the time from the date of first documented tumour response to the date of first documented disease progression or death due to underlying cancer. Patients with no event at the time of the analysis will be censored.
Time to Treatment Failure (TTF) | up to 36 months
  The Time to Treatment Failure will be defined as the time from the date of randomisation to the date of permanent study treatments discontinuation (any cause, including disease progression, treatment toxicity, adverse event, start of any new anticancer therapy, withdrawal of consent and death). Patients without treatment failure at the time of the analysis will be censored at the date of last tumour
Overall Survival (OS) | up to 36 months
  The Overall Survival will be defined as the time from the date of randomisation to the date of death due to any cause. Any patient not known to have died at the time of analysis will be censored based on the last recorded date on which the patient was known to be alive.
Quality of Life (QoL) | up to 36 months
  The Quality of Life will be assessed using the EORTC QLQ-C30 questionnaire.
Tolerance profile | up to 36 months
  The Tolerance profile will be described through the incidence and severity of drug-related AEs according to the Common Terminology Criteria for Adverse Events (CTCAE) (v5.0)

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Institut de cancérologie Strasbourg Europe, Strasbourg, Bas-Rhin
  - Centre Léon Bérard, Lyon, Rhône
  - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hôpital Cochin, Paris
  - CHU de Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - Institut Claudius Regaud - IUCT Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif